CLINICAL TRIAL: NCT00976833
Title: Standardized Rehabilitation for ICU Patients With Acute Respiratory Failure
Brief Title: Standardized Rehabilitation for Intensive Care Unit (ICU) Patients With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007879
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Failure
Keywords: Acute Respiratory Failure; Early ICU Mobility; Early Physical Therapy; Critical Care; Intensive Care; ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual Care
  Interventions: Other: Usual Care
- Standardized Rehabilitation (Other): Intervention arm to receive Standardized Rehabilitation Therapy
  Interventions: Other: Standardized Rehabilitation

INTERVENTIONS:
Other: Standardized Rehabilitation — 3 component Rehabilitation approach, Passive Range of Motion, Physical Therapy and Progressive Resistance Training
  Arms: Standardized Rehabilitation
Other: Usual Care — Usual Physical Therapy care
  Arms: Usual Care

SUMMARY:
Acute Respiratory Failure (ARF) requiring mechanical ventilation affects 1.1 million of the 4.4 million people admitted to United States Intensive Care Units (ICU) every year. Patients with ARF have an average ICU and hospital length of stay (LOS) of 8 and 15 days, respectively, with median hospital costs greater than $30,000 United States. Patients with ARF experience deconditioning, muscle weakness, joint contractures, dyspnea, depression, and reduced health-related quality of life, all of which may contribute to prolonged hospitalization and increased costs. Mechanistically, it is understood that patients with ARF demonstrate acute inflammation which may contribute to the above cited problems. While the investigators' research and that of others has shown that rehabilitation therapy can increase functional outcomes while lowering biomarkers of inflammation in the frail aged and other clinical populations, it is not known whether such rehabilitation therapy can result in improved functional capacity and functional performance and reduce inflammation in ARF patients. There is previous evidence for the feasibility and safety of rehabilitation therapy in ARF patients. Therefore, the investigators propose a two-arm, randomized trial in 326 patients with ARF to compare Standardized Rehabilitation Therapy initiated in the ICU and administered throughout the hospitalization versus usual care (control). Standardized Rehabilitation Therapy will consist of: passive range of motion, physical therapy and progressive resistance exercise (strength training). The regimen will be administered 7 days/week by a Mobility Team consisting of a critical care nurse, physical therapist and nursing assistant.

The investigators will determine whether standardized rehabilitation therapy will reduce hospital LOS, improve functional capacity and performance, improve quality of life, reduce inflammation and reduce hospital costs as compared to usual care.

This study's primary objective is to determine whether standardized rehabilitation therapy will decrease hospital length of stay.

Hypothesis: Compared to usual care, standardized rehabilitation therapy will reduce hospital length of stay for patients with Acute Respiratory Failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mechanically ventilated via an Endotracheal tube or Bipap
* Lung Injury

Exclusion Criteria:

* Previously enrolled in TARGET STUDY
* Inability to walk without assistance prior to acute ICU illness (use of a cane or walker not exclusion)
* Cognitive impairment prior to acute ICU illness (non-verbal)
* Acute stroke
* Body mass index (BMI) > 50
* Neuromuscular disease that could impair weaning
* Hip fracture, unstable cervical spine or pathological fracture
* Mechanically ventilated > 80 hours
* Current hospitalization or transferring hospital stay > 7 days
* Ineligible cancer treatment within the last 6 month
* Moribund
* Do Not Resuscitate(DNR)/Do Not Intubate(DNI) on admission
* Other Research Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine whether standardized rehabilitation therapy will decrease hospital length of stay. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Morris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gandotra S, Lovato J, Case D, Bakhru RN, Gibbs K, Berry M, Files DC, Morris PE. Physical Function Trajectories in Survivors of Acute Respiratory Failure. Ann Am Thorac Soc. 2019 Apr;16(4):471-477. doi: 10.1513/AnnalsATS.201806-375OC. PMID 30571923
- [Derived] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766